CLINICAL TRIAL: NCT04643353
Title: Use of Non-ablative Vaginal Erbium YAG Laser for the Treatment of Stress Urinary Incontinence.
Acronym: VELSUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Jan Deprest, MD, PhD, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S64486
Record Dates: First submitted 2020-11-18; First posted 2020-11-25 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-05

CONDITIONS: Urinary Incontinence,Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-ablative vaginal Erbium YAG laser treatment (Experimental): There are 3 visits where vaginal application of laser will be performed, with a 4-weeks interval. If needed, 3 extra laser applications can be added to the treatment (ie. with a maximum of 6 applications). Each application lasts around 15 minutes. The vaginal laser procedure will be performed in an outpatient setting, not requiring any specific preparation, analgesia or anesthesia, by one of two experienced operators.
  Laser therapy is performed using a 2940 nm VEL (SP Spectro, Fotona, Slovenia)with SMOOTH mode setting, which enables non-ablative, thermal-only operation). The parameters are selected based on extensive preclinical and clinical studies.
  Each laser treatment session consists of a full vaginal canal irradiation (using a 360° circular adapter), followed by additional irradiation of the prolapsed anterior wall (using a 90° angular adaptor) and concluded with irradiation of the vestibule area.
  Interventions: Device: Non-ablative vaginal Erbium YAG laser treatment
- Pelvic floor exercises (PFE) (Active Comparator): Standard PFE in Belgium are 9 sessions with a pelvic floor physiotherapist of choice, which can be extended by another 9 sessions, if clinically indicated. There are different strategies, though that will be on discretion of the physiotherapist. We will register the type of physiotherapy (standard (PFMT) versus assisted pelvic floor muscles training (APFMT)), number of completed sessions and duration of therapy. What is exactly done by the patient is registered as a variable.
  Interventions: Other: PFE

INTERVENTIONS:
Device: Non-ablative vaginal Erbium YAG laser treatment — Laser therapy is performed using a 2940 nm VEL (SP Spectro, Fotona, Slovenia) with SMOOTH mode setting, which enables non-ablative, thermal-only operation. The parameters are selected based on extensive preclinical and clinical studies.
  Arms: Non-ablative vaginal Erbium YAG laser treatment
Other: PFE — PFE will be prescribed as it is already implemented in clinical practice (i.e. up to 2x 9 sessions with a pelvic floor physiotherapist of choice). Type of physiotherapy, number of completed sessions and duration of therapy will be recorded.
  Arms: Pelvic floor exercises (PFE)

SUMMARY:
This is a single center, investigator initiated study, sponsored by the UZ Leuven, Leuven, Belgium; comparing laser treatment to pelvic floor exercises (PFE).

Women with symptomatic stress urinary incontinence who seek for a conservative treatment, with no history of previous incontinence-surgery will be randomised to either the laser-arm or the PFE-arm.

There are 3 visits (with a maximum of 6 visits) where vaginal application of laser will be performed, with a 4-weeks interval. Each application lasts around 15 minutes. The vaginal laser procedure will be performed in an outpatient setting, not requiring any specific preparation, analgesia or anesthesia, by one of two experienced operators.

The primary objective is to evaluate the effects of VEL treatment for the subjective cure or improvement of SUI.

The secondary objectives are to measure objective outcomes, to register any adverse events, and to determine for how long the effects of laser are sustained, with a maximum of two years.

ELIGIBILITY:
Inclusion Criteria:

* The presence of mild (score 1-2) to moderate (3-6) SUI with wish for treatment. The patient can have concomitant urge urinary incontinence (UUI), but that should not be the leading factor. Incontinence severity will be categorized by the four-level Sandvik severity index score (SIS). Scores are from 0 to 12. The higher the score, the more severe the urinary incontinence (mild=1-2, moderate= 3-6, severe=8-9, very severe=12).
* Voluntary informed consent

Exclusion Criteria:

* Any previous PFE-treatment in the last year for the same problem
* Previous surgery for incontinence or prolapse
* Severe (Sandvik SIS ≥8) SUI or insensible loss, high suspicion of intrinsic sphincter deficiency (ISD)
* Prolapse grade III or more
* Pregnancy
* Vaginal bleeding, injuries or infection in the treated area

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Primary outcome is the subjective success rate (cure or improvement) of SUI | 4 months after randomisation
  The tool used is the UDI-6 questionnaire. Converted UDI-6 scores range between 0 and 300. The "minimum important difference" is defined as a (MID)=11. In that score, cure is defined as answering "No" (0) to the question "Do you experience urine leakage related to physical activity, coughing or sneezing?".

SECONDARY OUTCOMES:
Assessment of overall urinary symptoms by means of the Urogenital Distress Inventory (UDI-6). | At every visit (ie. week 4, 8 and 12), end of initial treatment (ie. 4 months after randomisation), 6, 12 and 24 months after end of treatment
  The final UDI-6 score is calculated by adding all scores, and dividing the result to 6 to obtain a mean value which is in turn multiplied by 25 to obtain the scale score. The score varies from 0 to 100. The basic interpretation of the score is that the higher the score, the higher the disability . This questionnaire is available and validated in English , Dutch and French .
Assessment of the objective success rate by means of the cough stress test (CST). | At every visit (ie. week 4, 8 and 12), end of initial treatment (ie. 4 months after randomisation), 6, 12 and 24 months after end of treatment
  A working group of the International Continence Society (ICS) has developed instructions on the performance, interpretation and reporting of the CST in a standardized manner: the ICS-Uniform Cough Stress Test (ICS-UCST).
  For the ICS-UCST it is recommended that the patient is in a supine/lithotomy position with 200-400 mL of fluid in the bladder, which can be non-invasively assessed with a bladder scan. She coughs forcefully 1-4 times and the examiner directly visualizes the urethral meatus for the presence of leakage. Leakage of fluid from the urethral meatus coincident with/ simultaneous to the cough(s) is considered a positive test. If the test is negative (i.e, no leakage detected), then accessory stress testing such as repeating the test in the upright position should be considered.
Assessment of the rate of patient satisfaction by means of the Patient Global Impression of Improvement (PGI) | At every visit (ie. week 4, 8 and 12), end of initial treatment (ie. 4 months after randomisation), 6, 12 and 24 months after end of treatment
  5-point Likert scale (1=much worse, 2=worse, 3=same, 4=better, 5=much better)
Assessment of the degree of discomfort of the treatment procedure by the patient | At every visit (ie. week 4, 8 and 12), end of initial treatment (ie. 4 months after randomisation), 6, 12 and 24 months after end of treatment
  VAS-score (0-10cm, continuous scale)
Assessment of the longevity of the effect of laser therapy | At every visit (ie. week 4, 8 and 12), end of initial treatment (ie. 4 months after randomisation), 6, 12 and 24 months after end of treatment
  measured by the need for, and the timing for repeating the same, or initiating an alternative therapy.
Assessment of sexual function | At every visit (ie. week 4, 8 and 12), end of initial treatment (ie. 4 months after randomisation), 6, 12 and 24 months after end of treatment
  by means of the Pelvic Organ prolapse/Urinary Incontinence Sexual Questionnaire IUGA revised (PISQ-IR). The PISQ-IR is a questionnaire with twenty questions. Q1 is a dividing question on being sexually active or not. Not sexually active (NSA) women are referred to Q2-Q6. Sexually active (SA) women are asked to fill out Q7-Q20. The questionnaire for NSA women consists of five questions or 12 items. A higher score refers to a higher impact of the PFD on sexual functioning. The questionnaire for SA women consists of 14 questions wherein women with a partner have to fill out all 14, being 22 items. Women without partner can skip questions 13 and 14, filling out 19 items. A lower score refers to a lower impact of the PFD on sexual functioning. This questionnaire is available and validated in English, Dutch and French .
Assessment of treatment compliance in the PFE-group | At end of initial treatment (ie. 4 months after randomisation), 6, 12 and 24 months after end of treatmentAt every visit (ie. week 4, 8 and 12), end of initial treatment (ie. 4 months after randomisation), 6, 12 and 24
  Therefore we will monitor how many of the participants attended the PFE treatment complete all sessions with their physical therapist.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Deprest, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No